CLINICAL TRIAL: NCT06635369
Title: The Role of Taurine in Periodontitis and Aging: a Preliminary Study
Brief Title: Taurine in Periodontitis and Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Hadi Sayedyousef, Phd candidate, Istanbul Medipol University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1078
Record Dates: First submitted 2024-10-04; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Peridontal Disease; Aging
Keywords: Taurine; Periodontitis; Aging; Inflammation; TNF-α; SIRT1; Biomarker
MeSH Terms: conditions — Periodontitis; Inflammation

STUDY DESIGN:
Intervention Model Description: Participants are separated into four different groups. Young (25-44 years) with a healthy periodontium, young with periodontitis, old (≥65 years) with a healthy periodontium, and old with periodontitis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Young (25-44 years) with a healthy periodontium (Experimental)
  Interventions: Diagnostic Test: Periodontal Indices
- young (25-44 years) with Periodontitis (Experimental)
  Interventions: Diagnostic Test: Periodontal Indices
- Old (≥65 years) with a healthy periodontium (Experimental)
  Interventions: Diagnostic Test: Periodontal Indices
- Old (≥65 years) with Periodontitis (Experimental)
  Interventions: Diagnostic Test: Periodontal Indices

INTERVENTIONS:
Diagnostic Test: Periodontal Indices — Saliva, serum and periodontal indexes were obtained from patients
  Other Names: Salivary Flow Rate; TNF-α Levels; SIRT1 Levels; Taurine Levels

SUMMARY:
Aging leads to a decline in physiological functions and increases the risk of chronic diseases. Periodontitis is a chronic inflammatory disease that causes progressive destruction of the tissues supporting the teeth. Taurine, an amino acid with anti-inflammatory and antioxidant effects, might impact both periodontitis and aging. This study investigated taurine, SIRT1, and TNF-α levels in saliva and blood of 66 healthy people in different age groups, with or without periodontal disease. The findings showed that young people with healthy periodontal status had higher levels of taurine and SIRT1 compared to others. TNF-α, a marker of inflammation, was linked to the severity of periodontitis and may help identifying it in younger individuals. Overall, higher TNF-α levels are associated with periodontal inflammation, while taurine levels decrease with age-related inflammation.

ELIGIBILITY:
Exclusion Criteria:

* ages 18-25 or 45-64
* use of antibiotics, anti-inflammatory drugs, immunosuppressants, beta-blockers, calcium channel blockers, or anticoagulants within the last 6 months
* presence of diabetes, rheumatoid arthritis, or other systemic conditions such as cardiovascular, renal, hepatic, and neurodegenerative disorders
* pregnancy or lactation
* alcoholism
* smoking
* nonsurgical periodontal treatment in the past 6 months or surgical treatment in the past 12 months
* having less than 20 natural teeth, excluding third molars
* use of orthodontic appliances

Min Age: 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Taurine | 12 Weeks
  Taurine levels in saliva and serum were measured
SIRT1 | 12 Weeks
  SIRT1 levels in saliva and serum were measured
TNF-α | 12 Weeks
  TNF-α levels in saliva and serum were measured

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Unkapani, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to patients data privacy